CLINICAL TRIAL: NCT06406764
Title: A Randomized Controlled Trial Evaluating the Effect of Plyometric Training on Power, Speed, and Agility in Sport-active Boys With Different Biological Maturity
Brief Title: Effects of a Plyometric Training Program on Youths With Different Biological Maturity in Sport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Assistant professor, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FTK_2024_10
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Athletic Performance; Muscle Fatigue; Plyometric Exercise
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training (Experimental): Plyometric training program for 12 weeks.
  Interventions: Other: Plyometric training
- Control training (Active Comparator): Regular training program for 12 weeks.
  Interventions: Other: Control training

INTERVENTIONS:
Other: Plyometric training — Participants undergo a plyometric training program. The plyometric training consists of exercises in the horizontal, lateral, and vertical directions of movement. Exercises are progressively focused on maximal performance with short ground contact (<250 ms). The training sessions are twice per week.
  Arms: Plyometric training
Other: Control training — Participants continues their regular sports activities without additional plyometric training. The training sessions are twice per week.
  Arms: Control training

SUMMARY:
This randomized controlled trial aims to assess the effectiveness of a 12-week plyometric training regimen on improving power, speed, and agility among boys aged 10 to 18 years who are actively engaged in sports and exhibit differing levels of biological maturity. The study seeks to determine how maturation affects the responsiveness to the training program, potentially influencing future sports training approaches for young athletes.

DETAILED DESCRIPTION:
The main objective of this project is to assess the impact of a plyometric program on power, speed, agility, reactive strength index and stiffness in male athletes of different levels of maturation. The study takes the form of a short-term experiment (12 weeks), involving 30 young athletes with a minimum of two years of experience in systematic sports training. Participants are divided into an experimental group and a control group. The experimental group undergoes a 12-week plyometric training program, implemented twice a week within training sessions immediately following warm-ups. The control group engages in technical-tactical exercises. The program is developed by the authors of the research project based on current knowledge and requirements for creating an effective and safe plyometric program. Randomization is performed using a computer random generator. Participants undergo two testing sessions: one prior to the training intervention and the other one week after its completion. Age, height, weight, and body composition are measured using a personal scale with an integrated stadiometer. Tests include a 30-m sprint, countermovement jump, broad jump, unilateral triple jump, drop jump (reactive strength index), 20 submaximal vertical jumps (lower limb stiffness), BlazePod reaction test, and 505 agility test. The maturity status of the participants is evaluated using the Mirwald method and is used as a covariate in the subsequent statistical analysis. Findings of this research may provide crucial insights for targeted integration of plyometric methods during the developmental and maturation phases of young athletes.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 2 years of organized sports participation.
* Good health as confirmed by a pre-study medical screening.
* Signed informed consent from the legal representative and verbal assent from the participant.

Exclusion Criteria:

* Any serious lower limb injury in the past 6 months.
* Any current or historical mental health disorders.
* Any condition deemed by the medical screener as a contraindication to vigorous physical activity.

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Vertical jump height | 12 weeks
  The vertical jump is performed on AMTI OR6-7-1000 force platform (Advanced Mechanical Technology, Watertown, USA). Participants stand on the force platform in an upright position and on command, perform a maximum height jump with a countermovement and use of arms. Participants perform three attempts, with a 1-min rest between each. The best attempt is evaluated.
Broad jump distance | 12 weeks
  The distance in the broad jump is measured with a tape. Participants stand on a pre-marked line with legs approximately shoulder-width apart. From standing, they jump as far forward as possible using a countermovement and land on both feet. The landing spot closest to the starting line is considered for scoring. Participants perform two attempts, with the better attempt being recorded. There is a 1-min rest between attempts.
Unilateral triple jump length | 12 weeks
  The length of the unilateral triple jump test is measured with a tape. Participants start on one leg on a pre-marked line. Then using a countermovement from knee flexion, they perform a triple jump with the dominant and subsequently the non-dominant lower limb. After the final jump, they must land on both limbs and maintain their position at the landing spot for at least 2 seconds.

SECONDARY OUTCOMES:
Linear speed | 12 weeks
  A 20-m sprint test is used to assess linear speed. The final time is recorded using photoelectric cells (Brower Timing System, Draper, USA) with accuracy of 0.01 s. Photocells are placed at the start and 20-m mark. Participants start on command, with timing starting as soon as the player begins to move.
Agility test | 12 weeks
  For the 505 agility test, photoelectric cells (PR1aW, ALGE-TIMING, Lustenau, Austria) are used, placed at the 10-m mark. Cones are placed at the 0, 10, and 15-m marks. Participants sprint 10 meters and are instructed to reach maximum speed by the 10-m mark. At the 15-m mark, they perform a 180-degree turn and sprint back to the 10-m mark at maximum speed. Each participant have one attempt on the dominant and one attempt on the non-dominant leg for the 180-degree turn.
Reaction test | 12 weeks
  In the BlazePod reaction test (Play Coyotta, Tel Aviv, Israel), 5 sensors are placed parallel, 1 m apart from each other. The participant stand 3 m in front of the middle sensor. When any sensor lights up, the participant must press it as quickly as possible and return to the starting position, waiting for the next sensor to light up. Sensors light up in a random order. The test lasts after 10 attempts.
Lower limb stiffness | 12 weeks
  Lower limb stiffness is measured using the repeated submaximal jumps test (Optojump Next, Microgate, Italy). Participants perform 20 repeated jumps at a frequency of 2.5 Hz (mechanical metronome Wittner, Isny, Germany). Participants stand approximately shoulder-width apart with their hands on their sides throughout the test. Participants undergo three attempts with 2-min rest in between.
Reactive strength index | 12 weeks
  Reactive strength index is measured using the drop jump on AMTI OR6-7-1000 force platform (Advanced Mechanical Technology, Watertown, USA). Participants stand with feet shoulder-width apart on a platform 30 cm above the floor and have their hands on their sides. Then they step off the platform with one foot and upon landing, rebound as quickly as possible and with maximum effort. Reactive strength index is calculated from the ratio of jump height to the duration of contact with the platform.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Holik, Mgr, Principal Investigator — Palacky University, Faculty of Physical Culture
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw data will be made available.
Time Frame: The data will be available once the results are published in a scientific journal.
Access Criteria: For everybody.